CLINICAL TRIAL: NCT02291211
Title: Phase Ⅱ Study of S-1 Combined Cisplatin Hyperthermic Intraperitoneal Chemotherapy for Palliative Operation Gastric Cancer of Stage IV Limited Peritoneal Metastasis
Brief Title: S-1 Combined Cisplatin HIPEC for Palliative Operation Gastric Cancer of Stage IV Limited Peritoneal Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDCCC006
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-09

CONDITIONS: Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 plus cisplatin HIPEC (Experimental): 8 cycles of hyperthermic intraperitoneal chemotherapy (cisplatin) and S-1(oral) were performed after palliative operation gastric cancer of stage IV limited peritoneal metastasis. HIPEC was conducted in d1 and d3: Normal saline 2000ml-5000ml, Cisplatin 60mg/m^2, 43°C, 60min. every 3 weeks. S-1: 40-60mg/m^2 bid, days 1-14, every 3 weeks.Subjects should be given maximum 8 cycles, or progression/intolerance.
  Interventions: Drug: S-1 plus cisplatin HIPEC

INTERVENTIONS:
Drug: S-1 plus cisplatin HIPEC — Using cisplatin in HIPEC plus oral S-1
  Other Names: hyperthermic intraperitoneal chemoperfusion

SUMMARY:
This study is designed to investigate the efficacy of S-1 plus cisplatin hyperthermic intraperitoneal chemotherapy for advanced gastric patients of gastric cytoreductive surgery (CRS)

DETAILED DESCRIPTION:
This project is a single-center, open clinical observation the safety and efficacy that stage IV limited peritoneal metastasis of gastric cancer patients accept S-1 plus hyperthermic intraperitoneal chemotherapy . With advanced gastric patients of confined to the peritoneal after CRS as the research object, with progression-free survival and overall survival, adverse events as the end points.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 70 years old
* Patients with histologically confirmed gastric cancer (adenocarcinoma), stage IV (limited to the abdominal cavity), accpeted palliative cytoreductive surgery and no prior chemotherapy, biological therapy or targeted anti-cancer therapy, etc.
* The Eastern Cooperative Oncology Group (ECOG) status ≤ 2
* Having given written informed consent prior to any procedure related to the study
* Expected survival time ≥3 months

Exclusion Criteria:

* Known to have abdominal viscera metastasis of gastric cancer patients
* Inadequate hematopoietic function which is defined as below:

  * white blood cell (WBC) less than 3,500/mm^3
  * absolute neutrophil count (ANC) less than 1,500/mm^3
  * platelets less than 80,000/mm^3
* Inadequate hepatic or renal function which is defined as below:

  * serum bilirubin greater than 2 times the upper limit of normal range
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN if no demonstrable liver metastases or greater than 5 times the ULN in the presence of liver metastases
  * blood creatinine level greater than 1.5 times ULN,Creatinine clearance < 60ml/min
* Receiving a concomitant treatment with other fluoropyrimidine drug or flucytosine drug
* Women who is pregnant or lactating or fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period (Including male)
* Psychiatric disorder or symptom that makes participation of the patient difficult
* Myocardial infarction, existing serious or unstable angina, and patients with cardiac insufficiency in 6 months
* Severe complication(s), e.g., paresis of intestines, ileus, radiographically confirmed interstitial pneumonitis or pulmonary fibrosis, glomerulonephritis ,renal failure, poorly-controlled diabetes
* Known DPD deficiency
* Have the history of allograft transplantation
* Conducted the autologous bone marrow transplantation in 4 weeks
* Participate in other clinical trial before the start of this trial in 4 weeks
* Patient compliance is bad or researchers believe that patients are not suitable for this treatment
* Known to have active hepatitis patients
* HER-2-positive patients (ICH3+or FISH+)
* History of severe hypersensitivity reactions to the ingredients of S-1 or Cisplatin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
PFS: Progression Free Survival | 2 years
  from randomization to disease progression or death

SECONDARY OUTCOMES:
OS: Overall Survival | 5 years
  from randomization to death from any cause
Safety as measured by recording the subjects' Adverse Events from randomization to termination | 2 years
  Record the subjects' AEs from randomization to termination

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, Professor, Principal Investigator — Tang-Du Hospital
Locations (1):
- IEC of Insititution for National Drug Clinical Trials,Tangdu Hospital,Fourth Military Medical University, Xi'an, Shaanxi, China